CLINICAL TRIAL: NCT02897219
Title: Phase III Study of ASP1941 Double-blind, Parallel-group Study in Combination With Insulin in Patients With Type 1 Diabetes Mellitus
Brief Title: A Study of ASP1941 in Combination With Insulin in Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1941-CL-6002
Record Dates: First submitted 2016-07-27; First posted 2016-09-13 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: SGLT2 inhibitor; ASP1941; type 1 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — ipragliflozin; Convulsive Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 ASP1941 (Experimental): ASP1941 will be administered for 24 weeks under double blind conditions.
  Interventions: Drug: ipragliflozin; Other: Insulin Therapy
- Part 1 Placebo (Placebo Comparator): Placebo will be administered for 24 weeks under double blind conditions.
  Interventions: Drug: Placebo; Other: Insulin Therapy
- Part 2 ASP1941 (Experimental): ASP1941 will be administered for 28 weeks under open label conditions.
  Interventions: Drug: ipragliflozin; Other: Insulin Therapy

INTERVENTIONS:
Drug: ipragliflozin — Oral administration once daily
  Other Names: ASP1941
  Arms: Part 1 ASP1941; Part 2 ASP1941
Drug: Placebo — Oral administration once daily
  Arms: Part 1 Placebo
Other: Insulin Therapy — Continuous subcutaneous insulin infusion or multiple daily injections as standard of care

SUMMARY:
The objective of this study is to confirm efficacy of ASP1941 based on the changes in HbA1c and to assess its safety in subjects with type 1 diabetes mellitus receiving ASP1941 once daily in combination with insulin for 24 weeks. This study will also assess the safety/efficacy of long-term treatment (52 weeks).

DETAILED DESCRIPTION:
This study consists of two parts. In Part 1, ASP1941 or placebo will be administered orally in a blind manner. In Part 2, the long-term safety and efficacy of ASP1941 will be evaluated in patients who have participated in the study and completed the Part 1.

ELIGIBILITY:
Inclusion Criteria:

* The subject has been diagnosed with type 1 diabetes mellitus
* The subject has been receiving insulin therapy for the treatment of diabetes mellitus.
* The subject has not switched from an insulin product to another insulin product or switched between continuous subcutaneous insulin infusion (CSII) and multiple daily injections (MDI).
* The subject has an HbA1c value between 7.5% and 11.0% and the difference of HbA1c value is within ± 2.0%.
* The subject has a fasting blood C-peptide level < 0.6 ng/mL.
* The subject has a body mass index (BMI) between 20.0 kg/m2 and 35.0 kg/m2.

Exclusion Criteria:

* The subject has type 2 diabetes mellitus.
* The subject has participated in a clinical study or post marketing study of another drug or medical equipment within 12 weeks (84 days) before providing written informed consent, or is currently participating in such a study.
* The subject has received treatment with ASP1941 (ipragliflozin) or participated in a clinical study of ASP1941 (excluding subjects who discontinued before the investigational period).
* The subject participated in this study previously.
* The subject has received a hypoglycemic agent other than insulin or an α-glucosidase inhibitor.
* The subject has proliferative retinopathy (except for those who have undergone photocoagulation etc. and whose symptoms are stable).
* The subject has experienced severe hypoglycemia.
* The subject has experienced diabetic ketoacidosis.
* The subject has chronic disease that requires the continuous use of corticosteroids, immunosuppressants, etc.
* The subject has symptomatic urinary tract infection or symptomatic genital infection.
* The subject has a history of recurrent urinary tract infection or recurrent genital infection.
* The subject has a history of cerebral vascular attack, unstable angina, myocardial infarction, vascular intervention, or another serious heart disease.
* The subject has a concomitant malignant tumor or a history of malignant tumor
* The subject has a history of an allergy to ASP1941 (ipragliflozin) and/or similar drugs (drugs possessing SGLT2 inhibitory action).
* The subject has psychiatric disorder that is inappropriate for participation in the study.
* The subject has drug addiction or alcohol abuse.
* The subject has severe infection or serious trauma, or is perioperative.
* The subject has a history of medically significant renal disease such as renovascular occlusive disease, nephrectomy and/or renal transplant.
* The subject has any symptoms of dysuria, anuria, oliguria, or urinary retention.
* The subject has severe renal impairment or end-stage renal failure requiring dialysis.
* The subject has an Aspartate Aminotransferase and/or Alanine Aminotransferase value that exceeds 2 times, or a total bilirubin value that exceeds 1.5 times the upper limit of the reference range.
* The subject has uncontrolled severe hypertension.
* The subject has serious gastrointestinal disease or a history of operation for serious gastrointestinal disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2017-07-22 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | Baseline and Week 24 (end of treatment period 1)

SECONDARY OUTCOMES:
Change from baseline in HbA1c | Baseline and up to Week 56
Change from baseline in Fasting plasma glucose | Baseline and up to Week 56
Change from baseline in self-monitored blood glucose level | Baseline and up to Week 56
Change from baseline in leptin | Baseline and up to Week 52
Change from baseline in glycoalbumin | Baseline and up to Week 52
Change from baseline in adiponectin | Baseline and up to Week 52
Change from baseline in glucagon | Baseline and up to Week 52
Change from baseline in number of units of insulin administered concomitantly | Baseline and up to Week 56
  Comprehensively assessed by basal insulin daily dose, bolus insulin daily dose and total insulin daily dose.
Change from baseline in body weight | Baseline and up to Week 56
Change from baseline in waist circumference | Baseline and up to Week 52
Safety assessed by incidence of adverse events | Up to Week 56
Safety assessed by sitting blood pressure | Up to Week 56
Safety assessed by sitting pulse rate | Up to Week 56
Safety assessed by standard 12-lead electrocardiogram | Up to Week 56
Safety assessed by laboratory tests: Hematology | Up to Week 56
Safety assessed by laboratory tests: Biochemistry | Up to Week 56
Safety assessed by laboratory tests: Urinalysis | Up to Week 56

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (36):
- Japan (36):
  - Site JP00005, Aichi
  - Site JP00028, Aichi
  - Site JP00003, Chiba
  - Site JP00013, Chiba
  - Site JP00035, Chiba
  - Site JP00022, Fukuoka
  - Site JP00023, Fukuoka
  - Site JP00031, Fukuoka
  - Site JP00002, Gunma
  - Site JP00011, Gunma
  - Site JP00006, Hiroshima
  - Site JP00033, Hokkaido
  - Site JP00034, Hokkaido
  - Site JP00021, Hyōgo
  - Site JP00009, Ibaraki
  - Site JP00010, Ibaraki
  - Site JP00004, Kanagawa
  - Site JP00015, Kanagawa
  - Site JP00016, Kanagawa
  - Site JP00019, Mie
  - Site JP00008, Nagasaki
  - Site JP00024, Nagasaki
  - Site JP00025, Nagasaki
  - Site JP00032, Nagasaki
  - Site JP00026, Niigata
  - Site JP00020, Osaka
  - Site JP00029, Osaka
  - Site JP00036, Osaka
  - Site JP00012, Saitama
  - Site JP00017, Shizuoka
  - Site JP00018, Shizuoka
  - Site JP00001, Tochigi
  - Site JP00030, Tokushima
  - Site JP00014, Tokyo
  - Site JP00027, Toyama
  - Site JP00007, Yamaguchi

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/hcp/study.aspx?ID=308